CLINICAL TRIAL: NCT06473207
Title: Neuroprotective Effect of Remote Ischemic Post-conditioning in Out-of-hospital Cardiac Arrest : a Randomized Open Label Controlled Trial
Brief Title: Neuroprotective Effect of Remote Ischemic Post-conditioning in Out-of-hospital Cardiac Arrest
Acronym: RIPOST-CA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-CHITS-010; 2023-A02457-38 (Other: Id-RCB)
Record Dates: First submitted 2024-06-17; First posted 2024-06-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Remote ischemic conditioning; Out-of-hospital cardiac arrest; Neuroprotection; Cardiac arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic post-conditioning (RIPOST) (Experimental): Patients subjected to three sessions of RIPOST (within the 4 hours following cardiac arrest and then 12 and 24 hours after cardiac arrest)
  Interventions: Other: Remote ischemic post conditioning sessions
- Sham procedure (Sham Comparator): Patients subjected to three sessions of a sham procedure (within the 4 hours following cardiac arrest and then 12 and 24 hours after cardiac arrest)
  Interventions: Other: Sham sessions

INTERVENTIONS:
Other: Remote ischemic post conditioning sessions — Three sessions of RIPOST (within the 4 hours following cardiac arrest and then 12 and 24 hours after cardiac arrest), as follows: four cycles of cuff inflation to 200 mmHg for 5 min and then deflation to 0 mmHg for another 5 min (40 min total duration of the intervention), using an inflatable thigh tourniquet
  Other Names: RIPOST
  Arms: Remote ischemic post-conditioning (RIPOST)
Other: Sham sessions — Three sessions of a sham procedure (within the 4 hours following cardiac arrest and then 12 and 24 hours after cardiac arrest), as follows : application of a thigh tourniquet during 40 min without any inflation
  Other Names: Sham
  Arms: Sham procedure

SUMMARY:
Patients admitted to intensive care unit (ICU) following an out-of-hospital cardiac arrest (OHCA) have a high morbidity and mortality rate, primarily due to ischemia-reperfusion (I/R) syndrome leading to anoxic-ischemic brain injury. Despite current recommended advanced life support therapies, no specific treatment or procedure has yet been shown to improve the neurological outcome of such patients.

Remote ischemic post-conditioning (RIPOST) which usually consists of applying brief and repeated cycles of ischemia alternating with reperfusion by inflating and deflating a blood pressure cuff or a pneumatic tourniquet placed around a limb, is a promising strategy to protect organs against I/R injury, including brain. Regarding cardiac arrest, pre-clinical studies have demonstrated an improvement in neurological outcome in animal subjects treated with RIPOST after cardiopulmonary resuscitation.

The aim of our study is to demonstrate the benefit of early RIPOST in OHCA patients in reducing neurological injury and organ failure related to I/R syndrome.

DETAILED DESCRIPTION:
The RIPOST trial is a prospective, single-center, randomized, open-label, parallel group trial.

Patients with inclusion criteria will be randomized in two parallel groups:

* Experimental group: standard of care associated to 3 RIPOST sessions : one within the 4 hours following cardiac arrest, one 12 hours after cardiac arrest and one 24 hours after cardiac arrest. A RIPOST session = four cycles of cuff inflation to 200 mmHg for five minutes and then deflation to 0 mmHg for another five minutes, using an inflatable thigh tourniquet (total duration of the session = 40 minutes).
* Control group: standard of care associated to 3 sham sessions at inclusion, 24, and 48 hours after inclusion. A sham session = application of the thigh tourniquet during 40 minutes without any inflation.

Inclusion duration: 24 months

Patient participation duration: 3 months

Study duration: 27 months

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest with stable return of spontaneous circulation (ROSC > 20 minutes)
* Patient receiving invasive mechanical ventilation for coma (Glasgow score < 8)
* Availability of a lower limb without intravenous infusion or tension cuff positioned on it
* Randomization and application of the first session of the tested procedure within 4 hours after ROSC
* Consent of a next-of-kin or inclusion in emergency procedure

Exclusion criteria :

* Age < 18 y.o or pregnancy
* Patient unable to walk without assistance, unable to support himself properly without assistance, bedridden, incontinent and requiring nursing constant attention and care (corresponding to a mRS equal to 4 or 5)
* Interval between cardiac arrest and ROSC (no flow + low flow) estimated > 60 minutes
* Unwitnessed cardiac arrest with asystole as first rhythm
* In-hospital cardiac arrest
* Refractory cardiac arrest (no ROSC considered as stable)
* Cardiac arrest from traumatic, hemorrhage, stroke or hanging supposed origin
* Mean arterial pressure < 65mmHg persisting despite appropriate vascular filling and vasopressor and/or inotropic support
* Active uncontrolled bleeding
* Contraindication or not possible to use a pneumatic tourniquet on none of the two lower limbs (amputations, intravenous infusion positioned on both lower limbs, tourniquet size incompatible with patient morphology)
* Implementation of extracorporeal arteriovenous circulation for refractory cardiac arrest or refractory cardiogenic shock before inclusion
* Patient already included in this study
* Inclusion in another interventional study
* Judicial protection measure
* Patient without French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Neurofilament light chain (NFL) blood level evolution between 6 and 72 hours after cardiac arrest occurrence | 72 hours after out-of-hospital cardiac arrest occurrence
  Blood samples will be performed at 6 and 72 hours after cardiac arrest to monitor NFL level evolution and this evolution will be compared between both arms (RIPOST and sham groups)

SECONDARY OUTCOMES:
Sepsis organ failure assessment score (SOFA) | 72 hours after out-of-hospital cardiac arrest occurrence
  SOFA will be assessed at 24, 48 and 72 hours after cardiac arrest, and compared between both arms
Rate of patients with NFL peak level >500 pg/mL | 72 hours after out-of-hospital cardiac arrest occurrence
  Blood samples will be performed at 6, 24, 48 and 72 hours after cardiac arrest to monitor NFL peak level and the rate of patients who will present a NFL peak level > 500 pg/mL will be compared between both arms.
Neuron-specific enolase (NSE) blood level evolution between 6 and 72 hours after cardiac arrest occurrence | 72 hours after out-of-hospital cardiac arrest occurrence
  Blood samples will be performed at 6, 24, 48 and 72 hours after cardiac arrest to monitor NSE levels and their evolution will be compared between both arms (RIPOST and sham groups)
S100B protein (PS100B) blood level evolution between 6 and 72 hours after cardiac arrest occurrence | 72 hours after out-of-hospital cardiac arrest occurrence
  Blood samples will be performed at 6, 24, 48 and 72 hours after cardiac arrest to monitor PS100B levels and their evolution will be compared between both arms (RIPOST and sham groups)
ICU mortality rate from multi-organ failure and from neurological injury | At intensive care unit (ICU) discharge, up to 28 days
  Death mode at ICU discharge will be collected in both arms
Modified Rankin Scale (mRS) | 90 days after out-of-hospital cardiac arrest occurrence
  Modified Rankin Scale (mRS) will be assessed for both arms, at patient's ICU discharge and at day 90 after inclusion. This scales goes from 0 to 6, 0 corresponding to the absence of cognitive deficits and 6 to death.
Post out-of-hospital cardiac arrest event occurrence | 24 hours after out-of-hospital cardiac arrest occurrence
  Post out-of-hospital cardiac arrest event occurrence will be compared between both arms within the 24 hours following cardiac arrest. Events that will be considered are : unexpected cardiac arrest in ICU, iatrogenic events, limb ischemia, occlusive syndrome, digestive ischemia and thromboembolic complications.

CONTACTS AND LOCATIONS:
Overall Officials: Chelly Jonathan, MD, Study Director — Centre Hospitalier Intercommunal Toulon-La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon-La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho AFW, Chong J, Ong MEH, Hausenloy DJ. Remote Ischemic Conditioning in Emergency Medicine-Clinical Frontiers and Research Opportunities. Shock. 2020 Mar;53(3):269-276. doi: 10.1097/SHK.0000000000001362. PMID 32045394
- [Background] Kloner RA, Shi J, Dai W, Carreno J, Zhao L. Remote Ischemic Conditioning in Acute Myocardial Infarction and Shock States. J Cardiovasc Pharmacol Ther. 2020 Mar;25(2):103-109. doi: 10.1177/1074248419892603. Epub 2019 Dec 11. PMID 31823646
- [Background] Albrecht M, Meybohm P, Broch O, Zitta K, Hein M, Grasner JT, Renner J, Bein B, Gruenewald M. Evaluation of remote ischaemic post-conditioning in a pig model of cardiac arrest: A pilot study. Resuscitation. 2015 Aug;93:89-95. doi: 10.1016/j.resuscitation.2015.05.019. Epub 2015 Jun 4. PMID 26051813
- [Background] England TJ, Hedstrom A, O'Sullivan SE, Woodhouse L, Jackson B, Sprigg N, Bath PM. Remote Ischemic Conditioning After Stroke Trial 2: A Phase IIb Randomized Controlled Trial in Hyperacute Stroke. J Am Heart Assoc. 2019 Dec 3;8(23):e013572. doi: 10.1161/JAHA.119.013572. Epub 2019 Nov 21. PMID 31747864
- [Background] Moseby-Knappe M, Mattsson N, Nielsen N, Zetterberg H, Blennow K, Dankiewicz J, Dragancea I, Friberg H, Lilja G, Insel PS, Rylander C, Westhall E, Kjaergaard J, Wise MP, Hassager C, Kuiper MA, Stammet P, Wanscher MCJ, Wetterslev J, Erlinge D, Horn J, Pellis T, Cronberg T. Serum Neurofilament Light Chain for Prognosis of Outcome After Cardiac Arrest. JAMA Neurol. 2019 Jan 1;76(1):64-71. doi: 10.1001/jamaneurol.2018.3223. PMID 30383090